CLINICAL TRIAL: NCT03591302
Title: Total Lymphoid Irradiation, Anti-Thymocyte Globulin and Purified Donor CD34+ and T-cell Transfusion to Withdraw Immunosuppressive Drugs From Recipients of a Previous HLA Matched Living Donor Kidney Transplantation .
Brief Title: Delayed Blood Stem Transplantation in HLA Matched Kidney Transplant Recipients to Eliminate Immunosuppressive Drugs.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stephan Busque (Other)
Responsible Party: Sponsor-Investigator, Stephan Busque, Professor for Surgery, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46787
Record Dates: First submitted 2018-06-18; First posted 2018-07-19 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Immune Tolerance
Keywords: Kidney Transplantation; Blood Stem Cell Transplantation
MeSH Terms: interventions — Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: Total Lymphoid Irradiation, Anti-Thymocyte Globulin and Purified Donor CD34+ and T Cell Transfusion in previous HLA Matched Living Donor Kidney Transplantation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immune tolerance, Kidney transplantation (Experimental): Intervention: HLA matched living donor recipients of a functioning kidney transplant graft at one year will receive hematopoietic cell transplantation and Total lymphoid irradiation. The intervention is intended to induce immune tolerance such as to allow withdrawal of the immunosuppressive drugs. Immune tolerance is achieved through the development of donor/recipient mixed chimerism following combined kidney and hematopoietic stem cell transplantation from the living donor.
  Interventions: Biological: Hematopoietic cell transplantation; Radiation: Total Lymphoid irradiation

INTERVENTIONS:
Biological: Hematopoietic cell transplantation — Transplantation of hematopoietic stem cells from living donor.
Radiation: Total Lymphoid irradiation — Total lymphoid irradiation is used as part of the conditioning regimen for the hematopoietic stem cell transplant.

SUMMARY:
The study will determine whether patients with functioning Human Leukocyte Antigen (HLA) matched kidney transplants for at least one year and who want to discontinue immunosuppressive drugs can be treated with Total Lymphoid Irradiation (TLI) and rabbit Anti-Thymocyte Globulin (rATG) and an HLA matched donor hematopoietic progenitor cell infusion such that their drugs are successfully withdrawn while maintaining normal renal function.

DETAILED DESCRIPTION:
This is a single-center, open-label study in adult renal transplant patients.Twenty five patients with functioning HLA matched living donor kidney transplants will receive TLI, rATG and an infusion of cluster of differentiation (CD)34+ (Stem/Progenitor cells) selected granulocyte colony-stimulating factor (G-CSF) mobilized blood cells combined with CD3+ T cells (Stem/ Progenitor cells) from their transplant donors.Transplant recipients will have their maintenance Immunosuppressive drugs adjusted for four weeks before starting the TLI and ATG conditioning regimen. Mycophenolate Mofetil (MMF) will be maintained at 0.5 gm twice a day per day during this four week period during TLI and ATG treatments, and increased to 1 gram twice a day immediately after the completion of TLI at day 14.

MMF will be tapered starting 6 (six) months later. Tacrolimus levels will be targeted to blood trough levels of 4-6 ng/ml in the month before the start of the conditioning regimen. This target would be increased to 8-10 ng/ml at the start of the TLI and ATG conditioning regimen. At serial time points (1) graft function will be monitored. (2) chimerism will be measured in recipient white blood cell subsets, (3) protocol biopsies of the graft will be obtained. An attempt will be made to discontinue Tacrolimus at 12 months if (1) chimerism is detectable for least 180 days after the CD34+ and CD3+ cell infusion, (2) there is no Graft Versus Host Disease (GVHD), (3) there is stable graft function without clinical rejection episodes and (4) lack of histological rejection on protocol biopsies.

Recipients will be given the target dose of ≥ 8 x 10^6 CD 34 + cells/Kg and a dose of 5x10^6 CD3+ cells/Kg.The dose would be sequentially increased to 10, 15 and 25 x 10^6 CD3+ cells/Kg if fewer than 4 of 5 consecutive patients achieve whole blood chimerism of ≥ 30 % at 60 days. If 4 of 5 patients achieve this level of chimerism, then all subsequent enrolled patients will receive this dose.

ELIGIBILITY:
Inclusion Criteria:

1. All consenting adults of age 18 years and older with previous HLA matched sibling living donor renal transplants who still have their HLA- matched kidney donor available, and who have no history of acute or chronic rejection.
2. Patients who agree to participate in the study and sign an Informed Consent
3. The HLA-matched donor meets the Stanford Bone Marrow Transplant criteria for stem cell donation, agrees to participate and has signed an Informed Consent.
4. The pair is confirmed to be HLA-matched (2 haplo type match) as determined by the histocompatibility laboratory at Stanford.
5. Patients who have no known contraindication to the administration of rabbit ATG or radiation
6. Males and females of reproductive potential who agree to practice a reliable form of contraception for at least 18 months post transplant.

Exclusion Criteria:

1. Known allergy to ATG or a known allergy to rabbit proteins.
2. History of malignancy with the exception of non-melanoma skin malignancies.
3. Pregnant women or nursing mothers.
4. Serological evidence of HIV, Hepatitis B (HepBsAg+) or Hepatitis C infection.
5. Leukopenia (with a white blood cell count < 3000/mm3) or thrombocytopenia (platelet count < 100,000/mm3)
6. Previous history of acute or chronic rejection of the kidney transplant or recurrence of the original disease.
7. Screening kidney biopsy demonstrating acute or chronic rejection, recurrence of original disease or interstitial fibrosis/Tubular Atrophy (IF/TA) score greater than 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-09-13 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients no longer dependent on immunosuppressive drugs to maintain normal renal function. | six months to up to five years post stem cell transplant
  A patient will be considered no longer dependent if able to maintain normal renal function after coming off immunosuppressive medications.

SECONDARY OUTCOMES:
Percentage of patients experiencing biopsy proven rejection episodes requiring treatment requiring corticosteroids. | One year to five years
Percentage of patients experiencing graft loss. | One year to five years

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Md Strober, MD, Study Chair — Stanford University
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scandling JD, Busque S, Dejbakhsh-Jones S, Benike C, Millan MT, Shizuru JA, Hoppe RT, Lowsky R, Engleman EG, Strober S. Tolerance and chimerism after renal and hematopoietic-cell transplantation. N Engl J Med. 2008 Jan 24;358(4):362-8. doi: 10.1056/NEJMoa074191. PMID 18216356
- [Background] Scandling JD, Busque S, Shizuru JA, Engleman EG, Strober S. Induced immune tolerance for kidney transplantation. N Engl J Med. 2011 Oct 6;365(14):1359-60. doi: 10.1056/NEJMc1107841. No abstract available. PMID 21991976
- [Background] Scandling JD, Busque S, Dejbakhsh-Jones S, Benike C, Sarwal M, Millan MT, Shizuru JA, Lowsky R, Engleman EG, Strober S. Tolerance and withdrawal of immunosuppressive drugs in patients given kidney and hematopoietic cell transplants. Am J Transplant. 2012 May;12(5):1133-45. doi: 10.1111/j.1600-6143.2012.03992.x. Epub 2012 Mar 8. PMID 22405058
- [Background] Scandling JD, Busque S, Shizuru JA, Lowsky R, Hoppe R, Dejbakhsh-Jones S, Jensen K, Shori A, Strober JA, Lavori P, Turnbull BB, Engleman EG, Strober S. Chimerism, graft survival, and withdrawal of immunosuppressive drugs in HLA matched and mismatched patients after living donor kidney and hematopoietic cell transplantation. Am J Transplant. 2015 Mar;15(3):695-704. doi: 10.1111/ajt.13091. PMID 25693475
- [Background] Scandling JD, Busque S, Lowsky R, Shizuru J, Shori A, Engleman E, Jensen K, Strober S. Macrochimerism and clinical transplant tolerance. Hum Immunol. 2018 May;79(5):266-271. doi: 10.1016/j.humimm.2018.01.002. Epub 2018 Jan 9. PMID 29330112